CLINICAL TRIAL: NCT01321307
Title: Aphtostomatitis and Mucositis Treatment by Natural Herbal Formula (Sorend®)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: R&T Health Products Ltd. (Industry)
Responsible Party: Galit Avior, MD, Hillel Yaffe Medical Center
Other Study IDs: 91-2010-HYMC
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Aphtostomatitis; Mucositis
Keywords: Aphtostomatitis; Mucositis; Mouth sores; Natural; Herbal
MeSH Terms: conditions — Mucositis; Oral Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sorend: Group no. 1 shall receive Sorend following diagnosis of aphtostomatitis or mucositis.
- Sorend placebo: Group no. 2 shall receive Sorend placebo following diagnosis of aphtostomatitis or mucositis.

SUMMARY:
Sorend is a water-based formula, which contains carob, melissa and sage. Elder inhabitants of Israel are known to use carob extract to ease sores in the mouth, due to the tannins which create a complex with various proteins and polysaccharides, thus creating an impenetrable layer covering the sores, allowing spontaneous healing.

ELIGIBILITY:
Inclusion Criteria:

* Herpetic aphtomatitis
* Bacterial aphtostomatitis
* Viral aphtostomatitis
* Fungal aphtostomatitis

Exclusion Criteria:

* Oncology patients
* Systematic diseases (Colitis, Crohn, diabetes, Behcet)
* Pregnancy
* Arthritis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community population care
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2011-04

CONTACTS AND LOCATIONS:
Overall Officials: Galit Avior, MD, Principal Investigator — Hillel Yaffe Medical Center, Hadera, Israel
Locations (1):
- Hillel Yaffe MC, Otolaryngology - Head & Neck Surgery Unit, Hadera, Israel